CLINICAL TRIAL: NCT05580731
Title: Evaluation Study of Commercially Available Rapid Diagnostic Tests (RDTs) Detecting Antigen and Antibodies Against Dengue Virus
Brief Title: Evaluation Study of Dengue RDTs
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Sponsor
Other Study IDs: FE006B
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test: 5 different Rapid diagnostic test and Reference tests — Diagnostic test: 5 different Rapid diagnostic test and Reference tests

SUMMARY:
RT-PCR and virus isolation are considered gold standard for diagnosis of Dengue from blood during first few days of infection. Serological methods such as enzyme-linked immunosorbent assays (ELISA), confirms the presence of a recent or past infection with detection of NS1 antigen and anti-dengue antibodies. However, these methods are time-consuming and need significant laboratory infrastructure, including instrumentation, trained personnel and refrigeration for reagents. Hence, in areas where DENV is endemic, have limited resources and inadequate laboratory capacity to perform these tests, rapid diagnostic tests (RDTs) can be used for quick and simple screening. Recently various RDTs which detect Antigen (NS1) and Antibodies (IgM and IgG) in single format are widely available and in use, but the performance data are not available or not consistent from one study to another. Therefore, this study aims to evaluate the sensitivity and specificity of different RDTs that detect antigens and antibodies to Dengue viruses in one cassette during acute febrile stage thereby helping healthcare providers to decide on the best test.

DETAILED DESCRIPTION:
Dengue is an emerging infectious disease and is endemic to more than 100 tropical nations. It is a serious public health issue, with an estimated global incidence of > 100 million in 2016, a rise of almost 60% in age-standardized rates since 2006. While rising dengue infection rates affect all major regions of the world, the Asia-Pacific region is disproportionately affected by severe dengue, with rates 18 times higher in Southeast Asia than in the Americas. Climate change and globalization has facilitated the geographic spread of both the mosquito vector and the pathogen to previously unaffected areas, thereby increasing the number of people affected by dengue. Unfortunately, no specific antiviral medication and vaccine exists for Dengue. Hence, an accurate and early diagnosis is essential for proper and timely management and control of the disease in endemic regions. Dengue causes wide spectrum of disease. Primary dengue can range from sub clinical disease to flu-like symptoms. Although less common secondary dengue is associated with increased mortality and morbidity. Accurate, efficient, and rapid diagnosis of dengue in the acute stage is essential as a delay in diagnosis increases the risk of severe dengue and can lead to poor disease outcome. The most commonly used tests to diagnose acute dengue infection are commercial ELISA. Many Dengue RDTs came in rise and flooded the market in the past two decades due to the growing demand for point-of-care diagnostics. RDT is the easiest and most cost-effective method for diagnosis of this virus infection. It is user-friendly, requires no equipment and provide results faster than PCR and ELISA. Different format of Dengue RDTs are available in the market which can detect NS1, IgM and IgG. Detection of NS1, IgM and IgG in single RDT, not only detects primary dengue but also detects past dengue infection and can be helpful in disease prognosis. Many studies have been conducted previously focusing on individual markers of dengue RDTs and not the combined assessment of the test. This has significantly impeded healthcare providers to decide on deciding which overall tests is best to diagnose acute dengue and detects past dengue in a single test format. Hence, this study will aim to perform a head-to-head comparison of Dengue RDTs which detects antigen and antibodies in single test format currently in the market to diagnose acute dengue to help stakeholder decision making more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Have been obtained from patients presented with fever of < 1 week who have given consent for sample storage for further research purpose.
* Have minimum sample volume of 1 ml.
* Are non-haemolytic
* Have a limited number of freeze-thaw cycles (<3)
* Have been stored at or below -200C

Exclusion Criteria:

* Only samples that meet the inclusion criteria listed above will be selected for the study. Therefore, samples in the study site sample archives which do not meet these criteria will be excluded from the study.

Ages: 2 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at AKU research laboratory using leftover serum samples, which were archived for further research purposes for previous trial "Comparative study of commercially available typhoid point of care tests to benchmark current and emerging tools" conducted at AKU in 2020-2021. Precisely, the population is represented by children and adults (age 2-65) who presented with fever of 3-7 days duration. All patients from whom these samples were obtained have consented to store their sample at AKU and to use them for research on diagnostic tool for fever management.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity of each RDTs to detect acute dengue with 95% confidence intervals using ELISA as reference standard. | 7 months
  Point estimates of sensitivity and specificity, with 95% confidence intervals based on Wilson's score methods, will be calculated

SECONDARY OUTCOMES:
Estimates of operational characteristics of different RDTs, based on quantitative assessment including invalid rates | 7 months
  Rate of invalid runs: Percent of invalid runs per RDTs

CONTACTS AND LOCATIONS:
Overall Officials: Rumina Hasan, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided